CLINICAL TRIAL: NCT07014540
Title: Clinical Study on the Efficacy and Safety of Irinotecan Liposome Injection Combined With 5-FU/LV in the Treatment of Advanced Neuroendocrine Carcinoma
Brief Title: A Irinotecan Liposome Trial of in Advanced Neuroendocrine Carcinoma
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing GoBroad Hospital (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Ming Lu, Director, Beijing GoBroad Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DEY-NEC-BJ01
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Neuroendocrine Carcinomas (NEC)
MeSH Terms: conditions — Carcinoma, Neuroendocrine | interventions — Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Irinotecan hydrochloride liposome injection combined with 5-FU/LV therapy in a 2-week treatment cycle , until disease progresses or intolerable toxicity
  Interventions: Drug: Irinotecan Hydrochloride Liposome Injection; Drug: 5-FU; Drug: LV

INTERVENTIONS:
Drug: Irinotecan Hydrochloride Liposome Injection — Liposome irinotecan (70/50mg/m^2) will be administered by intravenous infusion on day 1 in a 2-week
Drug: 5-FU — 5-FU (2400mg/m^2) will be administered by continuous infusion for 46 hours in a 2-week
Drug: LV — LV (400mg/m^2) will be administered by intravenous infusion on day 1 in a 2-week

SUMMARY:
To explore the efficacy and safety of irinotecan liposome injection combined with 5-FU/LV in the treatment of advanced neuroendocrine carcinoma (NEC)

DETAILED DESCRIPTION:
1. Irinotecan hydrochloride liposome injection combined with 5-FU/LV therapy in a 2-week treatment cycle ,until disease progresses or intolerable toxicity

Drug: Liposome irinotecan(50-70mg/m^2) will be administered by intravenous infusion on day 1 in a 2-week treatment cycle

Drug: LV (400mg/m^2) will be administered by intravenous infusion on day 1 in a 2-week treatment cycle

Drug: 5-FU(2400mg/m^2) will be administered by continuous infusion for 46 hours on day 1 in a 2-week treatment cycle

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years
2. Advanced poorly differentiated neuroendocrine carcinoma diagnosed by histopathology, grade 3 (PD-EP-NEC, G3), after excluding the primary lesion in the lungs, cancers with unknown primary lesions are also allowed
3. Subjects who have failed at least the first-line standard treatment regimen in the past, recurrence within 6 months after the end of (new) adjuvant therapy is regarded as a failure of first-line treatment
4. Has not received irinotecan treatment
5. At least one measurable lesion，according to RECIST 1.1
6. ECOG 0~1
7. The expected survival ≥3 months
8. Having appropriate organ functions is defined as follows: those who need to complete hematological and blood biochemistry tests within 14 days before enrollment and meet the following conditions

   1. The absolute neutrophil count (ANC) was ≥1.5*10^9/L
   2. Hemoglobin ≥90g/dL
   3. Platelets (PLT) ≥100*10^9/L
   4. Total bilirubin <1.5 times the upper limit of normal value (ULN)
   5. Liver function Index (AST/ALT) chemical test <2.5 times the upper limit of normal value (ULN)
   6. Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance rate (CCr) ≥ 60mL/min, negative urine protein. For patients with urine protein ≥2+ at baseline, 24-hour urine collection should be conducted and the protein content in urine within 24 hours should be less than 1g
9. Patients with brain metastases enrolled in the group must meet the following conditions: (1) No clinical symptoms related to brain metastases and no need for systemic corticosteroids or anticonvulsant drugs for treatment; (2) No risk of cerebral hemorrhage
10. Male, female of childbearing age and their partners voluntarily adopted contraceptive measures considered effective by the researchers during the treatment and for at least three months after the last use of the study drug
11. Be able to understand and voluntarily sign the written informed consent form, which must be signed before carrying out the research procedures specified in any trial
12. Subjects fully understood and voluntarily participated in this study

Exclusion Criteria:

1. Within 28 days before the first treatment with the study drug, biological therapy, chemotherapy, surgical treatment, radiotherapy (PRRT requires 56 days), immunotherapy and other clinical study drug treatments (except placebo) were received; Small molecule drug treatment was received within 5 half-lives (for example, 6 days for everolimus and 10 days for sunitinib)
2. Adverse events caused by previous anti-tumor treatment (excluding alopecia) have not yet recovered (according to CTCAE. Version 5.0, with a severity level higher than level 1
3. Known active, uncontrollable or symptomatic central nervous system metastases, cancerous meningitis or leptomeningeal diseases suggested by clinical symptoms, cerebral edema and/or progressive tumor growth. Patients with a history of central nervous system metastasis or spinal cord compression, if they have received definite local treatments (such as radiotherapy, stereotactic surgery) and are clinically stable, and have stopped anticonvulsants and steroids for at least 4 weeks before enrollment, are eligible to be enrolled in this study
4. Known hemorrhagic constitution or disease
5. Patients with any severe and/or uncontrolled diseases

   1. Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months, and severe uncontrolled arrhythmia;
   2. Active or uncontrolled severe infections;
   3. Liver diseases such as liver cirrhosis, decompensated liver disease, and chronic hepatitis (i.e., positive for quantifiable HBV-DNA and/or HbsAg, and quantifiable HCV-RNA);
6. Hypertension that cannot be controlled by medication is defined as a systolic blood pressure of ≥140mmHg or a diastolic blood pressure of ≥90mmHg
7. There have been or are currently active ulcers of the stomach and duodenum, ulcerative colitis and other digestive tract diseases, or unresected digestive tract tumors with active bleeding, or other conditions that may cause digestive tract bleeding or perforation as determined by the researcher
8. Severe diarrhea (According to the NCI-CTCAE5.0 standard, grade 2 and above diarrhea: Compared with the baseline, the frequency of defecation increases by ≥4 times per day; Moderate to severe increase in the discharge from the stoma opening; Restrictions on daily living activities
9. Those who have a history of deep vein thrombosis, pulmonary embolism or other serious thromboembolism within 6 months before the first administration of the study drug
10. Subjects with serious injuries or non-healing wounds, or with unhealed fractures
11. Combined with uncontrollable systemic diseases (such as unstable angina pectoris, myocardial infarction, congestive heart failure, severe unstable ventricular arrhythmia, history of severe pericardial diseases and other cardiovascular diseases；uncontrollable hypertension, diabetes, etc.
12. Those who are known to be allergic or intolerant to therapeutic drugs or their excipients
13. Patients who participated in other interventional clinical studies simultaneously
14. Those with other malignant tumors requiring treatment
15. The researchers judged the patients who were not suitable to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | baseline up to approximately 2 months
  To evaluate the efficacy of anti-tumor

SECONDARY OUTCOMES:
overall survival (OS) | baseline up to approximately 6 months
  To evaluate the efficacy of anti-tumor
Progression-free survival (PFS) | baseline up to approximately 12 months
  To evaluate the efficacy of anti-tumor
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From the initiation of the first dose to 14 days
  To identify the incidence of AE and SAE in clinical trial

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing GoBroad Hospital, Beijing, Beijing Municipality, China